CLINICAL TRIAL: NCT04553926
Title: Lynparza Tablet (Olaparib) Regulatory Post-Marketing Surveillance
Brief Title: 'OLAP' (OLAparib Regulatory Post-marketing Surveillance)
Acronym: OLAP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00010
Record Dates: First submitted 2020-09-10; First posted 2020-09-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Breast Cancer; Prostate Cancer; Pancreatic Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objectives of this study are to assess safety and effectiveness of Lynparza tablet (olaparib, hereinafter "the study drug") in a real world setting in patients who are prescribed with the study drug according to the approved indications in South Korea

DETAILED DESCRIPTION:
Primary Objective: To assess the safety of the study drug for patients prescribed with the study drug under the approved indications in South Korea Secondary Objective: To assess effectiveness of the study drug for patients prescribed with the study drug under the approved indication in South Korea Exploratory Objective: To assess effectiveness of the study drug for ovarian cancer patients diagnosed as Homologous Recombination Deficiency (HRD) positive via locally available validated HRD test and prescribed with the study drug under the approved indication in South Korea

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for the study drug treatment according to the approved label in South Korea
2. Provision of signed and dated written informed consent by the patient or legally acceptable representative

Exclusion Criteria:

1. History of hypersensitivity to excipients of the study drug or to drugs with a similar chemical structure or class to the study drug
2. Prior exposure to any Polyadenosine 5'diphosphoribose polymerase (PARP) inhibitors, including the study drug
3. Pregnant and/or breast feeding
4. Current participation in any interventional trial
5. Other off-label indications according to the approved label

Ages: 19 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: On active study drug treatment according to the approved local label.
Sampling Method: Non-Probability Sample
Enrollment: 661 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events (AEs), serious AEs (SAEs), adverse drug reactions(ADRs), serious ADRs (SADRs), unexpected AEs/ADRs) | For about 1 year since the first dose of the study drug

SECONDARY OUTCOMES:
6-month real-world Progression free survival (rwPFS) | For about 1 year since the first dose of the study drug
  In this PMS, the secondary/pre-specified endpoint is not just PFS, but real-world PFS (rwPFS). That means the sponsor cannot claim investigator/patients to visit hospital for study assessment purposes.
  We, study sponsor, can only assess and record patient's disease progression status when patients visit hospital for their original follow-up. That's why we need further +50% duration for assessing rwPFS.

OTHER OUTCOMES:
1-year real-world Progression free survival (rwPFS) | For about 18 months since the first dose of the study drug
  for the exploratory objective, "In this PMS, the secondary/pre-specified endpoint is not just PFS, but real-world PFS (rwPFS). That means the sponsor cannot claim investigator/patients to visit hospital for study assessment purposes.
  We, study sponsor, can only assess and record patient's disease progression status when patients visit hospital for their original follow-up. That's why we need further +50% duration for assessing rwPFS.

CONTACTS AND LOCATIONS:
Locations (18):
- South Korea (18):
  - Research Site, Ansan
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Changwon
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Goyang
  - Research Site, Gunpo
  - Research Site, Hwaseong
  - Research Site, Ilsan
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Seongnam
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Uijeongbu-si
  - Research Site, Yangsan
  - Research Site, Yŏngin